CLINICAL TRIAL: NCT06493175
Title: The Application of Large Language Model in Emergency Chest Pain Triage
Acronym: ALERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Jinan Central Hospital (Other); Qingdao Municipal Hospital (Other); Tianjin Medical University General Hospital (Other); The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Tang Yida, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: M2023828
Record Dates: First submitted 2023-12-22; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Chest Pain
Keywords: large language model; Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large Language Model Diagnostic (Experimental): Patients interacted with the large-language model triage system MedGuide-V5 during the waiting period before or after routine triage in the emergency department. During this phase, MedGuide-V5 will automatically record data and metrics during communication with patients.
  Interventions: Diagnostic Test: Application of large language model in emergency chest pain triage.
- Routine diagnostic and therapeutic procedure (Active Comparator): After the artificial intelligence system evaluation, the patients will receive the diagnosis and treatment according to the normal procedure. The overall time of artificial triage, the triage of patients, and other data will be recorded. Patient visits should not be delayed by the use of artificial intelligence systems for evaluation.
  Interventions: Diagnostic Test: According to the normal procedures to receive medical treatment

INTERVENTIONS:
Diagnostic Test: Application of large language model in emergency chest pain triage. — The large language model MedGuide-V5 is able to quickly extract key information from a patients description, and by analyzing these descriptions, it provides physicians with a possible initial diagnosis to help them quickly prioritize the treatment of patients.
  Arms: Large Language Model Diagnostic
Diagnostic Test: According to the normal procedures to receive medical treatment — After the artificial intelligence system evaluation, the patients will receive the diagnosis and treatment according to the normal procedure. The overall time of artificial triage, the triage of patients, and other data will be recorded. Patient visits should not be delayed by the use of artificial intelligence systems for evaluation.
  Arms: Routine diagnostic and therapeutic procedure

SUMMARY:
This study will evaluate the accuracy and efficiency of large language model in emergency triage.

DETAILED DESCRIPTION:
The study is to evaluate the value of large language model in emergency triage, their accuracy and efficiency were evaluated and compared with traditional triage. To explore whether the model can effectively reduce the workload of medical staff, while improving the speed and quality of triage. In addition, the ability of the model to predict serious medical events such as acute heart events and strokes was evaluated. It also included surveys of patients; acceptance and satisfaction with the use of the artificial intelligence-assisted triage system. Analyze the economic benefits of adopting this technology, including cost saving and optimal allocation of resources.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with chest pain entered the emergency triage procedure.
2. patients aged 18 and above.

Exclusion Criteria:

1. Patients with severe cognitive impairment or inability to communicate.
2. There are patients who have been explicitly referred to specific departments (for example, some of the 120 transfer patients, who may go directly to the green channel) .
3. Patients with unstable vital signs .
4. Patients with potential medical problems.
5. Is participating in other clinical trials.
6. Failure to follow test procedures.
7. Those who refuse to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
The Diagnostic Accuracy Rate of MedGuide-V5 | through study completion, an average of 10 months
  To assess the consistency of the diagnosis of chest pain made by physicians with the assistance of large language models with the actual diagnosis made by patients after all examinations were completed.

SECONDARY OUTCOMES:
The Satisfaction of Medical Personnel | during evaluation
  To evaluate the satisfaction and acceptance of medical personnel with the use of large language models in assisting triage systems through methods such as questionnaire surveys. The name of this questionnaire is: Researcher Evaluation Form, with scores ranging from 1 to 10. The higher the score, the more helpful the large language model is to researchers.
Medical Personnel Treatment Plan Adjustment Rate | during evaluation
  The number of times medical personnel adjust treatment plans after receiving feedback from MedGuide V5's results and referring to the suggestions provided by the large language model.
Emergency Department Revisit Rate within 30 Days | during evaluation
  Evaluate the occurrence of patients revisiting the emergency department or being readmitted within 30 days after large language model-assisted triage and traditional triage.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No